CLINICAL TRIAL: NCT02240199
Title: Pregabalin and Lidocaine in Breast Cancer Surgery to Alter Neuropathic Pain (PLAN): A Pilot Trial
Brief Title: Perioperative Pregabalin and Lidocaine to Reduce Chronic Breast Cancer Pain
Acronym: PLAN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Hamilton Health Sciences Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PLAN14001
Record Dates: First submitted 2014-08-19; First posted 2014-09-15 (Estimated); Last update posted 2018-04-24 (Actual); Status verified 2016-12

CONDITIONS: Post-mastectomy Pain Syndrome; Chronic Post-surgical Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Lidocaine; Pregabalin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Pregabalin/Lidocaine (Experimental): Perioperative Pregabalin, Intraoperative Intravenous Lidocaine Infusion
  Interventions: Drug: Intraoperative Intravenous Lidocaine Infusion; Drug: Perioperative Pregabalin
- Pregabalin Placebo/Lidocaine (Active Comparator): Perioperative Pregabalin Placebo, Intraoperative Intravenous Lidocaine Infusion
  Interventions: Drug: Intraoperative Intravenous Lidocaine Infusion; Drug: Perioperative Pregabalin Placebo
- Pregabalin/Lidocaine Placebo (Active Comparator): Perioperative Pregabalin, Intraoperative Intravenous Lidocaine Placebo Infusion
  Interventions: Drug: Perioperative Pregabalin; Drug: Intraoperative Intravenous Lidocaine Placebo Infusion
- Pregabalin Placebo/Lidocaine Placebo (Placebo Comparator): Perioperative Pregabalin Placebo, Intraoperative Intravenous Lidocaine Placebo Infusion
  Interventions: Drug: Perioperative Pregabalin Placebo; Drug: Intraoperative Intravenous Lidocaine Placebo Infusion

INTERVENTIONS:
Drug: Intraoperative Intravenous Lidocaine Infusion — Lidocaine 1.5 mg/kg bolus with anesthesia induction followed by 2 mg/kg/hr infusion before the start of surgical incision and stopped at surgical closure.
  Other Names: Xylocaine
  Arms: Pregabalin Placebo/Lidocaine; Pregabalin/Lidocaine
Drug: Perioperative Pregabalin — Pregabalin 300 mg preoperatively (e.g. 2 hours prior to the start of surgery) and 75 mg twice a day for 9 days after surgery.
  Other Names: Lyrica
  Arms: Pregabalin/Lidocaine; Pregabalin/Lidocaine Placebo
Drug: Perioperative Pregabalin Placebo — Pregabalin placebo 300 mg preoperatively (e.g. 2 hours prior to the start of surgery) and 75 mg twice a day for 9 days after surgery.
  Arms: Pregabalin Placebo/Lidocaine; Pregabalin Placebo/Lidocaine Placebo
Drug: Intraoperative Intravenous Lidocaine Placebo Infusion — Lidocaine placebo 1.5 mg/kg bolus with anesthesia induction followed by 2 mg/kg/hr infusion before the start of surgical incision and stopped at surgical closure.
  Arms: Pregabalin Placebo/Lidocaine Placebo; Pregabalin/Lidocaine Placebo

SUMMARY:
Breast tissue and the areas surrounding the breast contain many small to medium-sized nerves. During surgery on the breast, these nerves can be inadvertently cut or damaged. Chemotherapy and radiotherapy after surgery worsen the injury experienced by these nerves. These nerves eventually become abnormal and provide pain signals to the brain well beyond the healing period after surgery. Patients with these abnormal nerves suffer from chronic pain in the breast area that persists for several years after surgery. Chronic pain is associated with a reduced quality of life, daily functioning, psychological distress, and contributes to excessive health care expenditures. There is encouraging data suggesting that an infusion of Lidocaine during surgery and Pregabalin given around the time of surgery can prevent the development of chronic pain after breast cancer surgery. A large randomized controlled trial is needed to determine the efficacy of these two interventions on reducing chronic pain after breast cancer surgery (e.g. within 3 months of surgery). A pilot trial is first needed to determine the feasibility of undertaking such a trial.

ELIGIBILITY:
Inclusion Criteria:

* female patients 18-75 years of age
* undergoing a unilateral or bilateral mastectomy or partial-mastectomy (breast conserving surgery), for prophylactic (e.g. family history or BRCA gene mutation) or belief of isolated (non-metastatic) cancerous lesions
* receiving a general anesthetic

Exclusion Criteria:

* previous breast surgery within six months of index surgery
* undergoing a DIEP (Deep Inferior Epigastric Perforator) flap procedure
* patient has chronic pain or a chronic pain syndrome for which they have taken 4 or more daily medications (i.e. opioids, anti-convulsants, anti-spasmodic, anti-depressants, anti-inflammatories) or routine pain intervention (i.e. nerve blocks) during the past 3 months
* documented hypersensitivity or allergy to pregabalin, gabapentin, or lidocaine
* history of ventricular tachycardia, ventricular fibrillation, or atrioventricular block ≥ type II
* history of congestive heart failure
* renal insufficiency with creatinine > 120 µmol/L
* known or previously documented cirrhosis
* pregnant
* unable to swallow study medications
* patient's surgeon believes patient is inappropriate for inclusion in trial
* unlikely to comply with follow-up (e.g. no fixed address, plans to move out of town)
* language difficulties that would impede valid completion of questionnaires
* patient requires gabapentin or pregabalin for a medical condition or has been taking gabapentin or pregabalin daily during the past 1 week

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2014-11; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Feasibility | 6 months
  The feasibility outcome will be measured by the rate of recruitment, compliance, percentage of patient's with complete follow-up and site resource requirements.

SECONDARY OUTCOMES:
Post-mastectomy pain syndrome | 6 months
Length of hospital stay | Total number of overnight stays spent in hospital continuously from the day of surgery until a maximum of 3 months post-operatively.
  Most breast cancer surgeries are day procedures, therefore length of hospital stay will be measured based on whether or not the patient was discharged from the hospital on the same day as surgery or if they were admitted and remained in hospital overnight.
Quality of Life | 3 months
Somatic Pre-occupation and Coping Scale | 3 months
Acute postoperative pain | Postoperative days 1-9

CONTACTS AND LOCATIONS:
Overall Officials: James S Khan, BHSc, MD, Study Director — Population Health Research Institute; P.J. Devereaux, MD, PhD, Principal Investigator — Population Health Research Institute
Locations (2):
- Canada (2):
  - Juravinski Hospital, Hamilton, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Khan JS, Hodgson N, Choi S, Reid S, Paul JE, Hong NJL, Holloway C, Busse JW, Gilron I, Buckley DN, McGillion M, Clarke H, Katz J, Mackey S, Avram R, Pohl K, Rao-Melacini P, Devereaux PJ. Perioperative Pregabalin and Intraoperative Lidocaine Infusion to Reduce Persistent Neuropathic Pain After Breast Cancer Surgery: A Multicenter, Factorial, Randomized, Controlled Pilot Trial. J Pain. 2019 Aug;20(8):980-993. doi: 10.1016/j.jpain.2019.02.010. Epub 2019 Mar 5. PMID 30844507